CLINICAL TRIAL: NCT01343797
Title: Glycemic and Insulinemic Index Determination of 2 Products: Fructilight® and A Fruit Fructo-Oligosaccharides in Sweet Matrix
Brief Title: Glycemic and Insulinemic Index Determination of Two Products: Fructilight® and A Fruit Fructo-Oligosaccharides in Sweet Matrix
Acronym: IGNUT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CRITT Bio-Industries (Other)
Collaborators: BioFortis (Other); NUTRITIS (Unknown)
Responsible Party: Françoise OUARNE, CRITT Bio-Industries
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IGNUT PEC10513
Record Dates: First submitted 2011-04-20; First posted 2011-04-28 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: Glycemic index; Insulinemic index; Fructo-oligosaccharide syrup; Fructose syrup; Aged between eighteen and fifty years old; BMI between nineteen and twenty five kg/m²; Non diabetic or pre-diabetic; Without liver, renal or gastro-intestinal disorder; Non-smoker
MeSH Terms: conditions — Glucose Intolerance; Digestive System Diseases

INTERVENTIONS:
Other: Glycemic and insulinemic index tests of a fruit fructose syrup and a fruit fructo-oligosaccharid syrup — One test with 65,5g of fruit (apple) extract sugar syrup with high fructose content in 250mL of water One test with 108,2g of peach purified sugar syrup with high fructo-oligosaccharid content in 250mL of water Three tests with the reference : 50g of anhydrous glucose in 250mL of water

SUMMARY:
The aim of the study is to determine glycemic and insulinemic index of 2 sweet syrups : FructiLight® and fruit Fructo-oligosaccharides in sweet matrix compared to glucose.

DETAILED DESCRIPTION:
12 male and female healthy adults are included in the study. During 5 separated visits subjects consume either 50 g of glucose in water (3 glucose response tests) or portion of syrup supply the equivalent of 50 g of glycaemic carbohydrates (2 syrup response tests).

Experimental sessions last 3 hours with 9 veinous and capillary blood taking. The experimental meals are served at t0 and are consumed between 12 and 15 minutes maximum. At time -5, 0, 15, 30, 45, 60, 90, 120 and 180 minutes, glucose is measured out on capillary blood and insulin is measured out on venous blood.

The glycemic index and Insulinemic index determination of the 2 syrups start by the calculation for each glycemia and insulinemia responses of the AUC over 120 min. The AUC(0-120min) is computed following the FAO recommendation (cf. FAO/WHO 1998), i.e. using the trapezoidal incremental method and not taking into account the area beneath the fasting concentration. then GI and II values expressed in percentage are calculated by dividing the AUC(0-120min) for test syrup products by the AUC(0-120min) for the glucose reference and multiplying by 100.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 50 years (limits included
* With a BMI between 19 and 25 kg/m² (limits included)
* Non-smoker
* Non-menopausal female with reliable contraception for two cycles before the beginning of the study and agreeing to keep it during the entire duration of the study
* Capable and willing to conform to the protocol and accepting to give his written informed consent
* Registered to Social Security System
* Accepting to be registered on the Volunteers in biomedical research file

After biological analysis, the subjects will be included on the following criteria :

* Fasting blood sugar level < 1,1 g/L
* Blood sugar level 120 minutes after 75g glucose intake < 1.4 g/L
* Complete blood count without significant clinically abnormality according to the investigator
* ASAT < 1,55 µkat/L
* ALAT < 1,7 µkat/L
* GGT < 2,55 µkat/L
* 45 < Creatinine < 104 µmol/L
* 1.7 < Urea < 8.3 mmol/L

Exclusion Criteria:

* Known food allergy, in particular to one of the tested products' components or to related products
* Personal history of hypercholesterolemia, high blood pressure, diabetes or glucose intolerance
* Renal insufficiency
* Liver disorders ongoing
* Gastrointestinal disorders, clinically significant according the investigator
* Use of medications which could affect lipidic or carbohydrate metabolism
* Disease or medication with impact on nutrients digestion and absorption
* Pregnant or breastfeeding women
* General anaesthetic in the month before the study
* Presenting a psychological or linguistic incapability to sign the informed consent
* Refusing to sign the informed consent
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros
* Impossible to contact in case of emergency
* Major or medical or surgical event with hospitalization in the last 3 months
* Taking part in an-other clinical trial or being in the exclusion period of a previous clinical trial

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Area Under the glycemia Curve over 120 min (AUC 0-120min) | 120 minutes after intake by test
  Syrup glycemic response compare to glucose glycemic response. Measure with glucometer at time 15, 30, 45, 60, 90, 120 (and 180 minutes) after the intake of 50g of glucose equivalent from the products (syrup or glucose). AUC(0-120min) calculation is computed following the FAO recommendation (cf. FAO/WHO 1998), i.e. using the trapezoidal incremental method and not taking into account the area beneath the fasting concentration.

SECONDARY OUTCOMES:
Area Under the insulinemia Curve over 120 min (AUC 0-120min) | 120 minutes after intake by test
  Syrup insulinemia response compare to glucose insulinemia response. Measure at time 15, 30, 45, 60, 90, 120 (and 180 minutes) after the intake of 50g of glucose equivalent from the products (syrup or glucose). AUC(0-120min) calculation is computed following the FAO recommendation (cf. FAO/WHO 1998), i.e. using the trapezoidal incremental method and not taking into account the area beneath the fasting concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Nantes, Pays de la Loire Region, France